CLINICAL TRIAL: NCT03825770
Title: A Pilot Randomized Controlled Trial of an Educational Program for Adults on Hemodialysis With Fatigue
Brief Title: Pilot Study of an Educational Program for Adults on Hemodialysis With Fatigue
Acronym: Fatigue-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Brenda Hemmelgarn, Department Head, Community Health Sciences, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1657
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Renal Dialysis; Fatigue; Rehabilitation; Quality of Life; Kidney Diseases
Keywords: Fatigue; Energy conservation; Rehabilitation; Occupational therapy; End-stage renal disease; Chronic kidney disease; Hemodialysis; Disability; Quality of life
MeSH Terms: conditions — Fatigue; Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: 1:1 pilot randomized controlled trial. Participants will be randomized to intervention (energy conservation education) or active control (general information about kidney disease).
Who Masked: Participant
Masking Description: Study participants will be blinded as to which educational program is the "active" treatment under study. Patient study materials and communications will only describe the study as being about an educational program for adults on hemodialysis with fatigue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The "PEP" Program (Experimental): The "PEP" (Personal Energy Planning) Program
  Interventions: Behavioral: The "PEP" (Personal Energy Planning) Program
- General Education (Active Comparator): General Education about Kidney Disease
  Interventions: Behavioral: General Education about Kidney Disease

INTERVENTIONS:
Behavioral: The "PEP" (Personal Energy Planning) Program — The PEP program is designed to teach people on dialysis with fatigue how to conserve energy during day-to-day tasks, and how to use energy conservation to accomplish their goals. The program is delivered over 7-9 weekly sessions. It consists of 2 educational web modules about energy conservation, and 5-7 goal-focused training sessions with a study clinician that utilize a problem-solving training approach known as the Cognitive Orientation to Occupational Performance (CO-OP) approach. Each program session lasts ~20-30 mins. Sessions are completed either in person during hemodialysis, or via telephone (based on patient preference). The program is administered by a trained study clinician (occupational therapist or nurse).
  Arms: The "PEP" Program
Behavioral: General Education about Kidney Disease — General education about kidney disease involves a review of information from the Kidney Foundation of Canada's patient handbooks "Living with Reduced Kidney Function" and "Living with Kidney Failure" (www.kidney.ca/manual) during 6-8 brief individual sessions with a trained study clinician (occupational therapist or nurse).The handbooks contains general information about managing kidney disease, addressing topics such as medication management, diet, and emotional well-being on dialysis. Sessions will take place either in person during hemodialysis, or via telephone (based on patient preference).
  Arms: General Education

SUMMARY:
Fatigue is a common and problematic symptom of end-stage renal disease (ESRD). The investigators have developed a new program, called the Personal Energy Planning (PEP) program, that teaches people with ESRD to manage fatigue by using energy conservation strategies during everyday life (eg. organization, prioritization, using good body postures and assistive tools). A large study is needed to test whether the program is helpful for people with ESRD. First, the investigators need to do a smaller-scale pilot study to help plan the large study. The main purposes of this pilot study are to see how many people with ESRD are willing and able to complete the PEP program, and to explore whether the program helps people feel less fatigued. The investigators plan to invite 40 people with ESRD from 4 dialysis units in Calgary, Alberta to participate. People with ESRD who report feeling unusually tired a lot of the time (using a symptom assessment tool completed every 2 months) will be asked to take part. Study participants will either do the PEP program, or another program (the control) that gives them general information about kidney disease. Participants will also be asked to complete questionnaires about fatigue before and after the study. The investigators will compare fatigue scores between the PEP program group and the control group, and record how many agree to take part in the study and complete all study activities. This pilot study will help the investigators plan next steps for research into the PEP program.

DETAILED DESCRIPTION:
BACKGROUND: Fatigue is one of the most common, disabling, and distressing symptoms experienced by people with end-stage renal disease (ESRD; kidney failure). There are currently few evidence-based treatment options to address fatigue in the ESRD population. Energy conservation education (ECE) is a rehabilitative approach shown to improve fatigue-related outcomes in other chronic disease populations, that has yet to be studied in people with ESRD. The investigators recently developed a novel ECE program for people with ESRD, conducted acceptability and usability testing, and showed improvements in fatigue and disability in single-case studies. A large randomized controlled trial (RCT) is now required to establish the efficacy of the PEP program, but additional feasibility information is first needed to design the definitive RCT.

OBJECTIVES:

1. To estimate the proportion of ESRD patients that are eligible for the RCT, will consent to participate, and will complete all study procedures
2. To identify the optimal primary outcome for the RCT and estimate the treatment effect size for RCT sample size calculations
3. To examine treatment fidelity to the PEP program among non-rehabilitation staff who undergo program administration training
4. To explore the effects of the PEP program on fatigue and disability at 3 months post-treatment

METHODS: Single-center, 1:1, parallel-arm pilot RCT. Adults on hemodialysis in Calgary at 4 dialysis units will be screened for eligibility. Prospective participants will be identified and approached by a clinical team member to assess their interest in the study. Interested patients will then be approached by a research team member to undergo informed consent and eligibility screening. Consenting participants will be randomized using a computer-generated randomization list and blocked randomization. Patients and outcome adjudicators will be blinded as to which is the treatment vs. control condition (blinding of providers is not feasible). Participants randomized to intervention will undergo the PEP energy conservation education program, consisting of two web modules and 4-7 sessions with a study clinician. Participants randomized to control will review the "Living with Kidney Disease" patient handbooks with a study clinician. Routine demographic and clinical data will be obtained at baseline, and the following measures will be administered to participants at baseline, mid-treatment, immediate post-treatment, and three months post-treatment: the Fatigue Severity Scale, Fatigue Impact Scale, Fatigue Management Questionnaire, Reintegration to Normal Living Index, and Canadian Occupational Performance Measure. A sample size of 40 patients (20 per arm) will provide an optimal estimate of treatment effect size for RCT sample size calculations, given 80% power, a small/medium effect size, and an attrition rate of ≤20%.

DATA ANALYSIS: The proportion of patients meeting each of the feasibility endpoints (eligibility, recruitment and attrition rates) will be calculated. Pre-to-post effect sizes will be calculated for all outcome measures used, and the outcome measure with the largest effect size will be chosen as the primary outcome for the RCT. Sample size calculations will then be made using the treatment effect size and variance from the pilot RCT data. Audio recordings of treatment sessions will be reviewed and rated using a Likert-scale rating system to estimate treatment fidelity. Effect sizes will also be calculated from pre-intervention to 3 months post-intervention.

IMPLICATIONS: Findings from this pilot RCT will help in the design of a robust RCT of the PEP program, which has the potential to improve fatigue management in the ESRD population.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* On chronic dialysis therapy for ≥3 months at time of recruitment
* Clinically and cognitively stable (able to provide informed consent)
* Scores an avg. of ≥4 on items 5, 7 , 8 and 9 of the Fatigue Severity Scale

Exclusion Criteria:

* Inadequate written and verbal English comprehension for study activities
* Plan in place to discontinue in-center hemodialysis at the participating center within 6 months of the time of recruitment (due to modality change, relocation, transplantation, or dialysis withdrawal)
* Resides in a nursing home facility
* Significant visual impairment (ie. unable to read size 14-pt font, Times New Roman)
* Scores >3 on Personal Health Questionnaire 2 (PHQ-2) depression screening tool

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Eligibility rate | From start to end of study screening (approximately 9 months)
  The proportion of patients screened who are eligible for the study
Recruitment rate | From start to end of study recruitment (approximately 9 months)
  The proportion of patients eligible for the study who consent to participate
Attrition rate | From start to end of study data collection (approximately 15 months)
  The proportion of consenting patients who withdraw from the study before completing all study activities

SECONDARY OUTCOMES:
Fatigue Severity Scale | From 1 week pre-intervention to 2 weeks mid-intervention, 1 week post-intervention, and 3 months post-intervention
  A 9-item self-report questionnaire which measures the severity of fatigue and its impact on activities and lifestyle
Fatigue Impact Scale | From 1 week pre-intervention to 2 weeks mid-intervention, 1 week post-intervention, and 3 months post-intervention
  A 21-item self-report questionnaire which assesses the effects of fatigue on physical, cognitive, and psychosocial functioning
Fatigue Management Questionnaire | From 1 week pre-intervention to 2 weeks mid-intervention, 1 week post-intervention, and 3 months post-intervention
  A 5-item self-report questionnaire which assesses self-perceived competence at fatigue management
Reintegration to Normal Living Index | From 1 week pre-intervention to 2 weeks mid-intervention, 1 week post-intervention, and 3 months post-intervention
  An 11-item self-report questionnaire which assesses the degree to which individuals who have experienced traumatic or incapacitating illness, achieve reintegration into normal social activities
Canadian Occupational Performance Measure | From 2 weeks mid-intervention to 1 week post-intervention, and 3 months post-intervention
  An outcome measure designed to capture a client's self-perception of performance in everyday living, over time

OTHER OUTCOMES:
Fidelity to treatment protocol | From start to end of study intervention (approximately 10 weeks per participant)
  Adherence to PEP program protocol by program administrators, measured by the Co-op Fidelity Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Brenda R Hemmelgarn, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- South Calgary Health Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murtagh FE, Addington-Hall J, Higginson IJ. The prevalence of symptoms in end-stage renal disease: a systematic review. Adv Chronic Kidney Dis. 2007 Jan;14(1):82-99. doi: 10.1053/j.ackd.2006.10.001. PMID 17200048
- [Background] Weisbord SD, Fried LF, Mor MK, Resnick AL, Unruh ML, Palevsky PM, Levenson DJ, Cooksey SH, Fine MJ, Kimmel PL, Arnold RM. Renal provider recognition of symptoms in patients on maintenance hemodialysis. Clin J Am Soc Nephrol. 2007 Sep;2(5):960-7. doi: 10.2215/CJN.00990207. Epub 2007 Aug 8. PMID 17702730
- [Background] Davison SN, Jhangri GS. Impact of pain and symptom burden on the health-related quality of life of hemodialysis patients. J Pain Symptom Manage. 2010 Mar;39(3):477-85. doi: 10.1016/j.jpainsymman.2009.08.008. PMID 20303025
- [Background] Ju A, Unruh M, Davison S, Dapueto J, Dew MA, Fluck R, Germain M, Jassal SV, Obrador G, O'Donoghue D, Josephson MA, Craig JC, Viecelli A, O'Lone E, Hanson CS, Manns B, Sautenet B, Howell M, Reddy B, Wilkie C, Rutherford C, Tong A; SONG-HD Fatigue Workshop Collaborators. Establishing a Core Outcome Measure for Fatigue in Patients on Hemodialysis: A Standardized Outcomes in Nephrology-Hemodialysis (SONG-HD) Consensus Workshop Report. Am J Kidney Dis. 2018 Jul;72(1):104-112. doi: 10.1053/j.ajkd.2017.12.018. Epub 2018 Mar 16. PMID 29551585
- [Background] Heiwe S, Clyne N, Dahlgren MA. Living with chronic renal failure: patients' experiences of their physical and functional capacity. Physiother Res Int. 2003;8(4):167-77. doi: 10.1002/pri.287. PMID 14730721
- [Background] Manns B, Hemmelgarn B, Lillie E, Dip SC, Cyr A, Gladish M, Large C, Silverman H, Toth B, Wolfs W, Laupacis A. Setting research priorities for patients on or nearing dialysis. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1813-21. doi: 10.2215/CJN.01610214. Epub 2014 May 15. PMID 24832095
- [Background] Artom M, Moss-Morris R, Caskey F, Chilcot J. Fatigue in advanced kidney disease. Kidney Int. 2014 Sep;86(3):497-505. doi: 10.1038/ki.2014.86. Epub 2014 Apr 2. PMID 24694985
- [Background] Mathiowetz VG, Finlayson ML, Matuska KM, Chen HY, Luo P. Randomized controlled trial of an energy conservation course for persons with multiple sclerosis. Mult Scler. 2005 Oct;11(5):592-601. doi: 10.1191/1352458505ms1198oa. PMID 16193899
- [Background] Finlayson M, Preissner K, Cho C, Plow M. Randomized trial of a teleconference-delivered fatigue management program for people with multiple sclerosis. Mult Scler. 2011 Sep;17(9):1130-40. doi: 10.1177/1352458511404272. Epub 2011 May 11. PMID 21561960
- [Background] Vanage SM, Gilbertson KK, Mathiowetz V. Effects of an energy conservation course on fatigue impact for persons with progressive multiple sclerosis. Am J Occup Ther. 2003 May-Jun;57(3):315-23. doi: 10.5014/ajot.57.3.315. PMID 12785670
- [Background] Kim YJ, Rogers JC, Raina KD, Callaway CW, Rittenberger JC, Leibold ML, Holm MB. Solving fatigue-related problems with cardiac arrest survivors living in the community. Resuscitation. 2017 Sep;118:70-74. doi: 10.1016/j.resuscitation.2017.07.005. Epub 2017 Jul 8. PMID 28698007
- [Background] Norberg EB, Lofgren B, Boman K, Wennberg P, Brannstrom M. A client-centred programme focusing energy conservation for people with heart failure. Scand J Occup Ther. 2017 Nov;24(6):455-467. doi: 10.1080/11038128.2016.1272631. Epub 2017 Jan 5. PMID 28052703
- [Background] Missiuna C, Mandich AD, Polatajko HJ, Malloy-Miller T. Cognitive orientation to daily occupational performance (CO-OP): part I--theoretical foundations. Phys Occup Ther Pediatr. 2001;20(2-3):69-81. PMID 11345513
- [Background] Polatajko HJ, Mandich AD, Missiuna C, Miller LT, Macnab JJ, Malloy-Miller T, Kinsella EA. Cognitive orientation to daily occupational performance (CO-OP): part III--the protocol in brief. Phys Occup Ther Pediatr. 2001;20(2-3):107-23. PMID 11345506
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Flachenecker P, Kumpfel T, Kallmann B, Gottschalk M, Grauer O, Rieckmann P, Trenkwalder C, Toyka KV. Fatigue in multiple sclerosis: a comparison of different rating scales and correlation to clinical parameters. Mult Scler. 2002 Dec;8(6):523-6. doi: 10.1191/1352458502ms839oa. PMID 12474995
- [Background] Learmonth YC, Dlugonski D, Pilutti LA, Sandroff BM, Klaren R, Motl RW. Psychometric properties of the Fatigue Severity Scale and the Modified Fatigue Impact Scale. J Neurol Sci. 2013 Aug 15;331(1-2):102-7. doi: 10.1016/j.jns.2013.05.023. Epub 2013 Jun 20. PMID 23791482
- [Background] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Carswell A, McColl MA, Baptiste S, Law M, Polatajko H, Pollock N. The Canadian Occupational Performance Measure: a research and clinical literature review. Can J Occup Ther. 2004 Oct;71(4):210-22. doi: 10.1177/000841740407100406. PMID 15586853
- [Background] Wood-Dauphinee SL, Opzoomer MA, Williams JI, Marchand B, Spitzer WO. Assessment of global function: The Reintegration to Normal Living Index. Arch Phys Med Rehabil. 1988 Aug;69(8):583-90. PMID 3408328
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476